CLINICAL TRIAL: NCT05135351
Title: A Pilot, Randomized, Double-blind, Placebo-controlled Study Using Prebiotics to Improve Gut Microbiome Diversity After Autologous Stem Cell Transplantation in Multiple Myeloma and Lymphoma: The PRIMAL Trial
Brief Title: Study Using Prebiotics to Improve Gut Microbiome Diversity After Autologous Stem Cell Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 0821-21-EP
Record Dates: First submitted 2021-11-18; First posted 2021-11-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Resistant Starch; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): resistant starch
  Interventions: Dietary Supplement: Resistant Starch
- Placebo (Placebo Comparator): maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Resistant Starch — A prebiotic nutritional supplement available at commercial grocery and health food stores. Specifically, we will be using Bob's Red Mill® potato starch.
  Arms: Treatment
Dietary Supplement: Maltodextrin — A starch commonly used as a placebo in prebiotic trials that is digested in the stomach and rapidly absorbed
  Arms: Placebo

SUMMARY:
Higher gut microbiome diversity has been associated with improved survival following autologous stem cell transplantation in multiple myeloma and lymphoma. This study hypothesises that prebiotic supplementation with resistant starch (RS) will improve gut microbiome diversity at time of stem cell engraftment. To test this, participants will either have RS or a placebo (maltodextrin) mixed into a food item of their choice for approximately 10 days prior to stem cell infusion and continue to the first day of neutrophil engraftment. The study will look at the difference in gut microbiome diversity between the RS and placebo arm collected at the engraftment timepoint, dietary evaluation to assess the impact of subject diet on microbiome response to intervention and serum sample collection to assess differences to gut permeability during transplant.

DETAILED DESCRIPTION:
Higher gut microbiome diversity has been associated with improved survival following autologous stem cell transplantation in multiple myeloma and lymphoma, but no strategies have been identified to date that specifically target the gut microbiome. The investigators hypothesize that prebiotic supplementation with resistant starch (RS) will improve gut microbiome diversity at time of stem cell engraftment.

To test this hypothesis, the study will be a randomized, double-blind, placebo-controlled trial of resistant starch versus placebo (maltodextrin) in participants with myeloma or lymphoma undergoing autologous stem cell transplantation. Thirty subjects will be randomized 1:1 to the RS or placebo arm, dosed at 20g daily for 3 days followed by an increased to 20g twice a day mixed into a food item of the participant's choice. The intervention will begin approximately 10 days prior to stem cell infusion and will continue until the first day of neutrophil engraftment (first day absolute neutrophil count >500) or approximately 30 days in total. Fecal samples will be collected at 4 timepoints for microbiome analysis: 1) at study enrollment 2) day of stem cell infusion 3) day +7 post auto transplant and 4) first day of engraftment defined as absolute neutrophil count >500 (approximately 10-14 days post-transplant).

The primary endpoint will be the difference in gut microbiome diversity between the RS and placebo arm collected at the engraftment timepoint. Secondary endpoints will include dietary evaluation to assess the impact of subject diet on microbiome response to intervention and serum sample collection to assess differences to gut permeability during transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent
2. Willing to comply with all study procedures and be available for the duration of the study
3. Has pathologically confirmed multiple myeloma, Non-Hodgkin lymphoma (DLBCL, mantle cell lymphoma, follicular lymphoma, or peripheral T-cell lymphoma), or Hodgkin lymphoma as determined on medical record review per standard of care transplant procedures (no tissue required for study)
4. Meeting a standard-of-care indication for autologous stem cell transplantation for the above diseases as determined by the investigator
5. Adult Individuals (male or female) at least 19 years of age
6. Meeting indications and recommended for first autologous stem cell transplantation by investigator

Exclusion Criteria:

1. History of bariatric surgery (i.e. gastric banding, sleeve gastrectomy, Roux-en-Y bypass), chronic gastrointestinal disease including chronic diarrheal illness or inflammatory bowel disease
2. Previous intolerance to fiber supplementation
3. Allergy or intolerance to potato starch or maltodextrin
4. Subject unwilling to comply with stool sample collection
5. Not suitable for study participation due to other reasons at the discretion of the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who adhere to >70% of scheduled doses of the intervention | 35 Days
  To understand the feasibility of the intervention in the proposed study population, the percentage of subjects who adhere to >70% of scheduled doses will be calculated

SECONDARY OUTCOMES:
Hospital Duration | 25 days
  To evaluate the duration of hospitalization according to intervention assignment by measuring time from stem cell transplant to day of discharge.
Rate of Neutropenic Fever | 25 Days
  To estimate the rate of neutropenic fever in the post-transplant setting according to intervention assignment. This is captured by cumulative incidence of neutropenic fever (ANC <1000, temperature >38.0⁰C) by day 30 according to intervention assignment
Rate of broad-spectrum antibiotic exposure | 25 Days
  To determine the rate of broad-spectrum antibiotic exposure during transplant according to intervention assignment by measuring the proportion of subjects receiving systemic antibiotic exposure.
Rate of gastrointestinal symptoms | 35 Days
  To determine the rate of gastrointestinal symptoms according to intervention assignment by using the patient-reported gastrointestinal symptom rating scale (GSRS.)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R D'Angelo, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No